CLINICAL TRIAL: NCT00725725
Title: A Multi-center, Double-blind, Fixed Dose Trial Examining the Efficacy and Safety of Org 25935 Versus Placebo as Augmentation to Cognitive Behavioral Therapy in Subjects With Panic Disorder
Brief Title: Org 25935 Versus Placebo as Augmentation to Cognitive-behavioral Therapy to Treat Panic Disorder (P05705)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05705; MK-8435-002 (Other: Merck Protocol); Org 172012 (Other: Organon Protocol)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy; N-methyl-N-(6-methoxy-1-phenyl-1,2,3,4-tetrahydronaphthalen-2-ylmethyl)aminomethylcarboxylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 mg Org 25935 (Experimental): Participants took a total of 3 doses of 4 mg Org 25935 prior to therapy sessions over a 2-week period.
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: Org 25935
- 12 mg Org 25935 (Experimental): Participants took a total of 3 doses of 12 mg Org 25935 prior to therapy sessions over a 2-week period.
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: Org 25935
- Placebo (Placebo Comparator): Participants took a total of 3 doses of placebo matched to Org 25935 prior to therapy sessions over a 2-week period.
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Participants underwent 5 weekly CBT session (sessions were 60-90 minutes in duration).
Drug: Org 25935 — 4 mg Org 25935 is given in tablet form, a single dose 2 hours prior to 3 CBT sessions. A total of 3 doses of trial medication is given over a 2-week period.
  Arms: 4 mg Org 25935
Drug: Org 25935 — 12 mg Org 25935 is given in tablet form, a single dose two hours prior to 3 CBT sessions. A total of 3 doses of trial medication is given over a two-week period.
  Arms: 12 mg Org 25935
Drug: Placebo — Placebo is given in tablet form, a single dose 2 hours prior to 3 CBT sessions. A total of 3 doses of trial medication is given over a 2-week period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Org 25935 vs. placebo given in combination with cognitive-behavioral therapy (CBT) to reduce the symptoms of panic disorder. It is hypothesized that treatment with Org 25935 at a dose of 4 mg or 12 mg will differ significantly from placebo with respect to the Panic Disorder Severity Scale (PDSS) total score over 3 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* is a male, or a female who is not of childbearing potential or who is non-pregnant, non-lactating and using a medically accepted method of contraception.
* is between the ages of 18 and 65, inclusive;
* signed written informed consent after the scope and nature of the investigation have been explained to them before Screening evaluations;
* is fluent in English;
* is diagnosed at Screening with current panic disorder, with or without agoraphobia;
* has a Clinical Global Impressions (CGI)-Severity score at Screening of >= 4 and <= 6;
* is currently taking no psychotropic medications or is able and willing to discontinue these medications prior to the first CBT session. Anti-depressant and anxiolytic medications are acceptable only if they are stabilized for at least 8 weeks prior to Screening;
* is able to complete all scheduled assessment and treatment visits and is willing to comply with the requirements of the study protocol.

Exclusion Criteria:

* is diagnosed with a primary Axis I disorder other than panic disorder;
* has a Screening Montgomery-Asberg Depression Rating Scale (MADRS) score of >= 35 (severe depression);
* has any history of bipolar disorder, psychotic disorder, or obsessive compulsive disorder;
* has a diagnosis of post traumatic stress disorder, eating disorder, or substance abuse or dependence (excluding nicotine) within the past six months;
* is known or suspected to have significant personality dysfunction that could, in the investigator's opinion, interfere with trial participation. Participants with known borderline or avoidant personality disorder are excluded;
* are at imminent risk of self-harm or harm to others, in the investigator's opinion based on clinical interview and responses provided on the Columbia Suicide Severity Rating Scale (C-SSRS). Participants must be excluded if they report suicidal ideation of Type 4 or 5 in the past 3 months or suicidal behavior in the past 12 months as measured by the C-SSRS at Screening;
* is currently a psychiatric inpatient or has been hospitalized for a psychiatric condition within the past year;
* has ever been diagnosed with organic brain syndrome, mental retardation, or other cognitive dysfunction that could interfere with their capacity to participate in CBT or to complete safety and efficacy assessments;
* has any history of head trauma causing ongoing cognitive impairment;
* has any history of seizures (apart from childhood febrile seizures);
* has an uncontrolled, unstable clinically significant medical condition (e.g., renal, endocrine, hepatic, respiratory, cardiovascular, hematologic, immunologic or cerebrovascular disease, or malignancy) that may interfere with the interpretation of safety and efficacy evaluations in the opinion of the investigator;
* has a clinically relevant visual disturbance, such as cataract, color blindness, macular degeneration, glaucoma, or retinal disease;
* has clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings at Screening that may interfere with the interpretation of safety or efficacy assessments in the opinion of the investigator;
* has a Corrected QT interval (QTc) value >450 milliseconds at Screening using Bazett's QTc formula;
* for females, has a positive result on serum pregnancy test (at Screening), or plan to become pregnant during the course of the trial;
* has a positive urine drug or alcohol breath test at Screening, unless the positive finding can be accounted for by documented prescription use;
* is unable or unwilling to comply with the investigator's instructions regarding drug and alcohol use during the trial period;
* has a history of sensitivity/idiosyncrasy to glutamatergic drugs or chemically related compounds or excipients which may be employed in the trial or to any other unknown drug used in the past;
* are receiving concurrent psychotherapy for the treatment of panic disorder [general supportive psychotherapy is acceptable if therapy was initiated at least 3 months prior to Screening] or have received a prior adequate trial of CBT for panic disorder;
* has been exposed to an investigational drug within 6 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-07-23 (Actual); Primary Completion 2010-04-23 (Actual); Study Completion 2010-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Nations KR, Smits JA, Tolin DF, Rothbaum BO, Hofmann SG, Tart CD, Lee A, Schipper J, Sjogren M, Xue D, Szegedi A, Otto MW. Evaluation of the glycine transporter inhibitor Org 25935 as augmentation to cognitive-behavioral therapy for panic disorder: a multicenter, randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2012 May;73(5):647-53. doi: 10.4088/JCP.11m07081. Epub 2012 Feb 21. PMID 22394471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult (18 to 65 years of age) male and female participants with a diagnosis of current panic disorder (PD; with or without agoraphobia [AGP]) were recruited.
Period: Overall Study
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Started | 14 | 15 | 17
Treated | 11 | 15 | 14
Completed | 10 | 11 | 12
Not Completed | 4 | 4 | 5
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 17 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (9.9) | 36.4 (8.9) | 32.8 (10.8) | 34.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 13 | 31
  Male | 5 | 6 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Panic Disorder Severity Scale (PDSS) Score From Baseline to End-of-Treatment (EOT)
Description: The mean change in PDSS score from baseline (Screening) to EOT (Day 36) was calculated for each arm. The PDSS is a 7-item clinician-rated scale that assesses multiple dimensions of panic disorder severity (e.g., frequency of panic attacks). Each item is scored on a 5-point Likert scale (0 to 4) with the total score ranging from a minimum of 0 to a maximum of 28 (higher scores indicate greater panic disorder severity).
Time Frame: Screening and Day 36
Population: The Intent-to-Treat (ITT) population consisted of all participants who received ≥1 dose of double-blind study medication and had PDSS assessments at Screening and EOT.
Measure: Mean (Standard Deviation); unit: PDSS Score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 13
PDSS Score
  Screening | 11.5 (1.51) | 15.8 (4.00) | 17.1 (3.99)
  EOT (Placebo n=12) | 5.3 (1.49) | 7.6 (4.62) | 6.6 (4.29)
  EOT - Screening (Placebo n=12) | -6.2 (2.15) | -8.2 (4.49) | -10.4 (4.23)
Statistical Analysis 1: Comparison: 4 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.3934, Mixed Models Analysis; Mean Difference (Final Values) = 1.5299, 95% CI 2-sided [-2.0781 to 5.1380]
Statistical Analysis 2: Comparison: 12 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.3515, Mixed Models Analysis; Mean Difference (Final Values) = 1.2667, 95% CI 2-sided [-1.4665 to 4.0000]

2. Secondary Outcome: Change in PDSS Score From Baseline to Visit 4
Description: The mean change in PDSS score from baseline (Screening) to Visit 4 (Day 22) was calculated for each arm. The PDSS is a 7-item clinician-rated scale that assesses multiple dimensions of panic disorder severity (e.g., frequency of panic attacks). Each item is scored on a 5-point Likert scale (0 to 4) with the total score ranging from a minimum of 0 to a maximum of 28 (higher scores indicate greater panic disorder severity).
Time Frame: Screening and Visit 4 (Day 22)
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and PDSS scores at Screening and Visit 4.
Measure: Mean (Standard Deviation); unit: PDSS Score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 13
PDSS Score
  Screening | 11.5 (1.51) | 15.8 (4.00) | 17.1 (3.99)
  Visit 4 (4 mg O n= 9; 12 mg O n=12) | 7.1 (4.08) | 10.5 (4.56) | 12.2 (4.00)
  Visit 4 - Screening (4 mg O n= 9; 12 mg O n=12) | -4.2 (3.70) | -5.3 (4.03) | -4.9 (4.52)
Statistical Analysis 1: Comparison: 4 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.3597, Mixed Models Analysis; Mean Difference (Final Values) = -1.8246, 95% CI 2-sided [-5.8307 to 2.1815]
Statistical Analysis 2: Comparison: 12 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.7770, Mixed Models Analysis; Mean Difference (Final Values) = -0.4414, 95% CI 2-sided [-3.5952 to 2.7124]

3. Secondary Outcome: Change in PDSS Score From Baseline to Follow-Up
Description: The mean change in PDSS score from baseline (Screening) to Follow-Up (Day 59) was calculated for each arm. The PDSS is a 7-item clinician-rated scale that assesses multiple dimensions of panic disorder severity (e.g., frequency of panic attacks). Each item is scored on a 5-point Likert scale (0 to 4) with the total score ranging from a minimum of 0 to a maximum of 28 (higher scores indicate greater panic disorder severity).
Time Frame: Screening and Follow-Up (Day 59)
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had PDSS scores at Screening and Follow-Up.
Measure: Mean (Standard Deviation); unit: PDSS Score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 13
PDSS Score
  Screening | 11.5 (1.51) | 15.8 (4.00) | 17.1 (3.99)
  Follow-Up (12 mg O, Placebo n=12) | 4.8 (2.20) | 7.4 (5.85) | 5.3 (4.56)
  Follow-Up - Screening (12 mg O, Placebo n=12) | -6.7 (2.54) | -8.3 (5.80) | -11.7 (4.23)
Statistical Analysis 1: Comparison: 4 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.2683, Mixed Models Analysis; Mean Difference (Final Values) = 2.3356, 95% CI 2-sided [-1.8933 to 6.5644]
Statistical Analysis 2: Comparison: 12 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.0844, Mixed Models Analysis; Mean Difference (Final Values) = 3.1317, 95% CI 2-sided [-0.4518 to 6.7152]

4. Secondary Outcome: Structured Clinical Interview for DSM-IV-TR Axis 1 Disorders, Patient Edition With Psychotic Screen (SCID-I/P With Psy Screen) Score at Screening
Description: The SCID-I/P with Psy Screen, Panic Disorder Module was used to score participants' PD (with [w] or without [w/o] AGP) as being current (full criteria for the disorder met), in full remission (IFR) [there are no longer any symptoms or signs of the disorder, but it is still clinically relevant to note the disorder], or in partial remission (IPR) [full criteria for the disorder were previously met, but currently only some of the symptoms or signs of the disorder remain] at baseline (Screening). The SCID-I/P is a diagnostic exam used to assess for Axis-1 mental disorders.
Time Frame: Screening
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had SCID-I/P with Psy Screen scores at Screening.
Measure: Number; unit: Participants
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 13
Participants
  PD w AGP: Current | 9 | 12 | 12
  PD w/o AGP: Current | 1 | 2 | 1

5. Secondary Outcome: SCID-I/P With Psy Screen Score at EOT
Description: The SCID-I/P with Psy Screen, Panic Disorder Module, was used to score participants' PD (w or w/o AP) as being current (full criteria for the disorder are met), IFR (there are no longer any symptoms or signs of the disorder, but it is still clinically relevant to note the disorder), or IPR (full criteria for the disorder were previously met, but currently only some of the symptoms or signs of the disorder remain) at EOT (Day 36). The SCID-I/P is a diagnostic exam used to assess for Axis-1 mental disorders.
Time Frame: Day 36
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had SCID-I/P with Psy Screen scores at EOT.
Measure: Number; unit: Participants
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 13 | 12
Participants
  PD w AGP: Current | 3 | 4 | 6
  PD w AGP: IFR | 0 | 1 | 0
  PD w AGP: IPR | 4 | 4 | 5
  PD w/o AGP: Current | 1 | 3 | 0
  PD w/o AGP: IFR | 0 | 0 | 1
  PD w/o AGP: IPR | 2 | 1 | 0

6. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) Score
Description: The mean change in CGI-S score from baseline (Screening) to EOT (Day 36) was calculated for each arm. The CGI-S is a clinician-rated instrument used to assess global severity of general anxiety symptoms. The instrument consists of a 7-point scale that the clinician uses to rate the severity of the patient's illness, from 1 (normal, not at all ill) to 7 (extremely ill).
Time Frame: Screening and Day 36
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had CGI-S scores at Screening and EOT.
Measure: Mean (Standard Deviation); unit: CGI-S Score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 13
CGI-S Score
  Screening | 4.0 (0.0) | 4.6 (0.74) | 4.8 (0.83)
  EOT (Placebo n=12) | 2.8 (0.42) | 3.1 (0.92) | 3.0 (1.13)
  EOT - Screening (Placebo n=12) | -1.2 (0.42) | -1.6 (0.85) | -1.8 (0.97)

7. Secondary Outcome: Change in Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A) Score
Description: The mean change in SIGH-A score from baseline (Screening) to EOT (Day 36) was calculated for each arm. The SIGH-A is a 14-item scale to assess anxiety in a clinical population. Each item is scored on a 5-point Likert scale (0 to 4) with the total score ranging from a minimum of zero to a maximum of 56 (higher scores indicate greater anxiety severity).
Time Frame: Screening and Day 36
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had SIGH-A scores at Screening and EOT.
Measure: Mean (Standard Deviation); unit: SIGH-A Score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 13
SIGH-A Score
  Screening | 17.2 (8.42) | 14.3 (6.37) | 14.6 (9.14)
  EOT (12 mg O n=13; Placebo n=12) | 9.7 (7.21) | 10.0 (6.43) | 8.5 (6.96)
  EOT - Screening (12 mg O n=13; Placebo n=12) | -7.5 (7.37) | -3.8 (5.97) | -6.4 (7.62)
Statistical Analysis 1: Comparison: 4 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.8894, Mixed Models Analysis; Mean Difference (Final Values) = 0.3456, 95% CI 2-sided [-4.6211 to 5.3124]
Statistical Analysis 2: Comparison: 12 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.3765, Mixed Models Analysis; Mean Difference (Final Values) = 2.0417, 95% CI 2-sided [-2.5526 to 6.6360]

8. Secondary Outcome: Change in Anxiety Sensitivity Index (ASI) Score
Description: The mean change in ASI score from baseline (Screening) to EOT (Day 36) was calculated for each arm. The ASI is a 16-item self-report questionnaire that assesses fear of anxiety sensations. Each item is scored on a 5-point Likert scale (0 to 4) with total score ranging from a minimum of 0 to a maximum of 64 (higher scores indicate greater fear of anxiety sensations).
Time Frame: Screening and Day 36
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had ASI scores at Screening and EOT.
Measure: Mean (Standard Deviation); unit: ASI Score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 12
ASI Score
  Screening | 31.1 (9.92) | 37.1 (9.56) | 37.5 (12.91)
  EOT (12 mg O n=13) | 20.1 (10.29) | 26.3 (10.56) | 24.8 (13.95)
  EOT - Screening (Placebo n=11) | -11.0 (10.23) | -10.8 (14.48) | -13.8 (13.58)
Statistical Analysis 1: Comparison: 4 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.8073, Mixed Models Analysis; Mean Difference (Final Values) = -1.2502, 95% CI 2-sided [-11.4963 to 8.9958]
Statistical Analysis 2: Comparison: 12 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.6610, Mixed Models Analysis; Mean Difference (Final Values) = 2.0291, 95% CI 2-sided [-7.2132 to 11.2714]

9. Secondary Outcome: Change in Montgomery-Asberg Rating Scale for Depression (MADRS) Score
Description: The mean change in MADRS score from baseline (Screening) to EOT (Day 36) was calculated for each arm. The MADRS is a 10-item clinical-administered scale designed to assess severity of depression. Each item is rated from 0 to 6, with total score ranging from 0 to 60 (higher MADRS scores indicate more severe depression).
Time Frame: Screening and Day 36
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had MADRS scores at Screening and EOT.
Measure: Mean (Standard Deviation); unit: MADRS score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 13
MADRS score
  Screening | 12.4 (8.03) | 11.1 (6.38) | 14.2 (9.20)
  EOT (12 mg O n=13, Placebo n=12) | 6.6 (4.33) | 7.0 (6.98) | 6.3 (5.12)
  EOT - Screening (12 mg O n=13, Placebo n=12) | -5.8 (6.76) | -4.2 (5.06) | -7.8 (8.53)
Statistical Analysis 1: Comparison: 4 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.7895, Mixed Models Analysis; Mean Difference (Final Values) = 0.7296, 95% CI 2-sided [-4.7291 to 6.1883]
Statistical Analysis 2: Comparison: 12 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.5488, Mixed Models Analysis; Mean Difference (Final Values) = 1.5260, 95% CI 2-sided [-3.5495 to 6.6015]

10. Secondary Outcome: Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Score
Description: The mean change in Q-LES-Q score from baseline (Screening) to EOT (Day 36) was calculated for each arm. The Q-LES-Q is a self-report questionnaire rating 16 aspects of quality of life, including physical health and mood. Scores range from 0 ("very poor") to 5 ("very good"), with total score ranging from 0 to 80 (higher O-LES-Q scores indicate greater quality of life).
Time Frame: Screening and Day 36
Population: The ITT population consisted of all participants who received ≥1 dose of double-blind study medication and had Q-LES-Q scores at Screening and EOT.
Measure: Mean (Standard Deviation); unit: Q-LES-Q Score
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 10 | 14 | 12
Q-LES-Q Score
  Screening | 49.8 (6.20) | 47.2 (8.88) | 45.3 (11.63)
  EOT (12 mg O n=11) | 56.6 (3.20) | 50.5 (9.32) | 55.3 (7.69)
  EOT - Screening (12 mg O n=11, Placebo n=11) | 6.8 (5.39) | 3.7 (5.06) | 10.8 (11.79)
Statistical Analysis 1: Comparison: 4 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.6516, Mixed Models Analysis; Mean Difference (Final Values) = -1.2766, 95% CI 2-sided [-6.9269 to 4.3738]
Statistical Analysis 2: Comparison: 12 mg Org 25935 vs Placebo; Test type: Superiority or Other; p = 0.0256, Mixed Models Analysis; Mean Difference (Final Values) = -6.1867, 95% CI 2-sided [-11.5864 to -0.7869]

11. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: The number of participants experiencing one or more AEs throughout the study period was determined. An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 59 days
Population: All treated participants are included in the safety analysis.
Measure: Number; unit: Participants
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 11 | 15 | 14
Participants | 8 | 12 | 5

12. Secondary Outcome: Number of Participants Discontinuing Study Therapy Due to AEs
Description: The number of participants withdrawing from study treatment during the treatment period was determined. An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 2 weeks
Population: All treated participants are included in the safety analysis.
Measure: Number; unit: Participants
Arm/Group | 4 mg Org 25935 | 12 mg Org 25935 | Placebo
Number analyzed (Participants) | 11 | 15 | 14
Participants | 1 | 3 | 1

ADVERSE EVENTS:
Time Frame: Up to 59 days
Groups:
- Org 25935 4 mg: Participants took a total of 3 doses of 4 mg Org 25935 prior to therapy sessions over a 2-week period.
- Org 25935 12 mg: Participants took a total of 3 doses of 12 mg Org 25935 prior to therapy sessions over a 2-week period.
Arm/Group | Org 25935 4 mg | Org 25935 12 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 8/11 | 12/15 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Org 25935 4 mg (N=11) | Org 25935 12 mg (N=15) | Placebo (N=14)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (4) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (3)
Mydriasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (3) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Visual brightness (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 1 (2)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 7 (13) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Derealisation (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0)
Dissociation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No